CLINICAL TRIAL: NCT02322541
Title: Dietary Absorption of Garlic Metabolites Following Garlic Consumption
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was suspended due to additional time needed for method development.
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS48
Record Dates: First submitted 2014-12-08; First posted 2014-12-23 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Focus is Understanding Absorption of Garlic Metabolites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Time Course (Experimental): Measurement of garlic metabolites over 24 hours following garlic intervention.
  Interventions: Other: Garlic Intervention

INTERVENTIONS:
Other: Garlic Intervention — Participants will consume an Allium-free controlled diet for 3 days. On the 4th day, they will consume a test meal containing garlic followed by blood and urine collections for 10 hours. On the 5th day, participants will have a fasting blood and urine collection.

SUMMARY:
The study will consist of a single 5-day dietary treatment period. Subjects will consume an Allium-free diet for 3 days. Alliums are vegetables such as garlic, onions, chives, shallots, and leeks. On day 4, subjects will consume a breakfast consisting of garlic and will then provide blood and urine samples for 10 hours, and on the following morning.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of age 25 to 75 years at beginning of study
* BMI between 18.5 and 30 kg/m2
* Fasting glucose < 126 mg/dl
* Blood pressure < 160/100 (controlled with certain medications)
* Fasting total blood cholesterol < 280 mg/dl
* Fasting triglycerides < 300 mg/dl

Exclusion Criteria:

* Younger than 25 years old or older than 75 years old
* Use of blood-thinning medications such as Coumadin (warfarin), Dicumarol (dicumarol), or Miradon (anisindione)
* Presence of kidney disease, liver disease, gout, certain cancers, thyroid disease, gastrointestinal, other metabolic diseases or malabsorption syndromes.
* Have been pregnant during the previous 12 months, are currently pregnant or lactating, or plan to become pregnant during the study
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanolamine, ephedrine, caffeine) during and for at least 6 months prior to the start of the study or a history of a surgical intervention for obesity
* Active cardiovascular disease (such as a heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within the last three months, stroke, or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in the past six months).
* Use of any tobacco products in past 6 months
* Unwillingness to abstain from herbal supplements for two weeks prior to the study and during the study
* Known (self-reported) allergy or adverse reaction to garlic
* Inability to tolerate garlic
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past twelve months and/or current acute treatment or rehabilitation program for these problems (Long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Allyl methyl sulfide | 24 hour
  Metabolite will be analyzed in blood and urine.
N-acetyl allylcysteine sulfoxide | 24 hour
  Metabolite will be analyzed in blood and urine.
N-acetyl-S-trans-1-propenylcysteine sulfoxide | 24 hour
  Metabolite will be analyzed in blood and urine.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States